CLINICAL TRIAL: NCT06842680
Title: Evaluating the Effectiveness of an Ultraprocessed Food Warning Label in Chile
Brief Title: Testing Ultraprocessed Food Labels in Chile
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Instituto de Nutrición y Tecnología de los Alimentos (Other); Bloomberg Philanthropies (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 24-2896b
Record Dates: First submitted 2025-02-18; First posted 2025-02-24 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-04

CONDITIONS: Diet, Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator)
  Interventions: Behavioral: Control
- Ultraprocessed warning label (Experimental)
  Interventions: Behavioral: Ultraprocessed warning label

INTERVENTIONS:
Behavioral: Control — Products do not carry ultraprocessed warning label. To match the current Chilean legislation, products carry octagonal nutrient labels when applicable.
  Arms: Control
Behavioral: Ultraprocessed warning label — Products carry ultraprocessed warning label. To match the current Chilean legislation, products carry octagonal nutrient labels when applicable.
  Arms: Ultraprocessed warning label

SUMMARY:
The goal of this experiment is to examine the effects of a warning label signaling that a product is ultraprocessed among a sample of Chilean parents. The main questions this experiment aims to answer are:

Do ultraprocessed warning labels on their own impact product purchase intentions?

Do ultraprocessed warning labels impact product purchase intentions in the presence of nutrient warning labels?

Do ultraprocessed warning labels help more consumers identify ultraprocessed foods?

Participants will be randomly assigned to a control arm or an ultraprocessed warning label arm. In both arms, products will carry nutrient warning labels, which are Chile's current policy. Participants will see three similar products, all of which will be ultraprocessed: one not high in any nutrients of concern, one high in sodium, and one high in sodium and saturated fat. For each product, participants will rate their purchase intentions and indicate whether they believe the product to be ultraprocessed. Researchers will compare results across arms.

DETAILED DESCRIPTION:
Participants will complete an online randomized experiment programmed in Qualtrics. After providing informed consent, participants will be randomly assigned to one of two arms: control (i.e., no ultraprocessed warning label) arm or ultraprocessed warning label arm. In both arms, products will carry nutrient warning labels, which are Chile's current policy.

In random order, participants will see three similar mock bags of potato chips. All products seen will be ultraprocessed, and thus carry an ultraprocessed warning label in the ultraprocessed warning label arm. Additionally, one of the products will not be high in any nutrients of concern, one product will be high in sodium, and one product will be high in sodium and saturated fat. For each product, participants will rate their purchase intentions, perceived healthfulness, and indicate whether they believe the product to be ultraprocessed.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Parent or guardian of child between 2-14 years old who has never been diagnosed with diabetes, high blood sugar, pre-diabetes or insulin resistance
* Residing in Chile

Exclusion Criteria:

* Less than 18 years old
* Not parent or guardian of child between 2-14 years old who has never been diagnosed with diabetes, high blood sugar, pre-diabetes or insulin resistance
* Not residing in Chile

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3645 (Actual)
Dates: Start 2025-07-14 (Actual); Primary Completion 2025-08-31 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
Purchase intentions, mean score | During exposure to intervention (i.e., study stimuli), assessed during one-time online 10-minute survey.
  How likely the participant would be to buy products will be measured by survey. Response options will be on a 5-point scale from "very unlikely" (coded as 1) to "very likely" (coded as 5), with higher scores representing a higher likelihood of buying products.
Correct identification of products as ultraprocessed | During exposure to intervention (i.e., study stimuli), assessed during one-time online 10-minute survey.
  Correct identification of products as ultraprocessed will be measured by survey. Response will be coded in a dichotomous 0-1 range, where 1 indicates that the participant correctly identified the products as ultraprocessed and 0 indicates that the participant did not correctly identify the products as ultraprocessed.

SECONDARY OUTCOMES:
Perceived product healthfulness, mean score | During exposure to intervention (i.e., study stimuli), assessed during one-time online 10-minute survey.
  How good or bad it would be to consume the product every day will be measured by survey. Response options will be on a 5-point scale from "very bad" (coded as 1) to "very good" (coded as 5), with higher scores representing a higher perceived product healthfulness.

CONTACTS AND LOCATIONS:
Overall Officials: Aline D'Angelo Campos, MPP, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- The University of North Carolina at Chapel Hill's Gillings School of Global Public Health, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
The Study Protocol and Statistical Analysis Plan will be shared prior to data collection. After data collection and analysis, a de-identified version of individual participant data and the analytic code will be shared through the Open Science Framework (OSF).
Supporting Information: Study Protocol, SAP
Time Frame: The Study Protocol and statistical analysis plan will be available by March 2025 (prior to data collection). A de-identified version of the data collected and analytic code used will become available after data collection and analysis and will remain available indefinitely.
Access Criteria: Open access.
URL: https://osf.io/

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-04-10): https://cdn.clinicaltrials.gov/large-docs/80/NCT06842680/Prot_SAP_000.pdf